CLINICAL TRIAL: NCT06365203
Title: Comparative Study of Through Knee Amputation Versus Above Knee Amputation Regarding Infection Rate and Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Adly Omar, Resident doctor at vascular surgery department at Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Through knee amputation
Record Dates: First submitted 2024-03-22; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Amputation of Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Through knee amputation (Active Comparator): Through knee amputation
  Interventions: Procedure: Through knee amputation; Procedure: Above knee Amputation
- Above knee Amputation (Active Comparator): Above knee Amputation
  Interventions: Procedure: Through knee amputation; Procedure: Above knee Amputation

INTERVENTIONS:
Procedure: Through knee amputation — Amputation Technique
Procedure: Above knee Amputation — Amputation Technique

SUMMARY:
The aim of this study is to search and compare outcomes of through knee amputation (TKA) and above knee amputation (AKA) in terms of Technique ,wound healing ,infection rate , function and ambulation

DETAILED DESCRIPTION:
Severe peripheral arterial disease with or without comorbid diabetes mellitus accounts for the majority of patients requiring major lower extremity amputations.

There is also an association between major extremity amputation and lower socio-economic status, attributed to lifestyle and comorbidities, living and working conditions, psychosocial factors, and access to affordable healthcare.

With a transfemoral prosthesis, the amputee weight bears through their ischial tuberosity which can cause discomfort when standing or ambulating. These challenges have been associated with greater abandonment of prosthesis use. An often over looked alternative within amputation surgery is through knee amputation (TKA), which currently comprises less than 5% of all major lower extremity amputations.

Compared with AKA, TKA is a less traumatic procedure with little disruption to thigh muscles, articular cartilage, menisci, and bone (especially with Knee Disarticulation), which in turn reduces post-operative infection and formation of bone spurs.

In contrast, AKA can also provide additional problems. Due to a shorter lever length of the residuum, the unilateral transfemoral amputee requires three times more energy to ambulate with a prosthetic limb compared with a unilateral transtibial amputee.

Among vascular surgeons, TKA is similarly rarely performed. Fear of poor wound healing and potential stump breakdown in longer soft tissue flaps needed to cover epicondyles of the distal femur are possible preconceived misconceptions. Historically, outcomes after TKA are acceptable, but scarce vascular literature exists reporting contemporary outcomes of TKA.

ELIGIBILITY:
Inclusion Criteria:

* Critical limb ischemia with sever infection with no role For BKA
* Acute late or total ischemia SFA with poor
* popliteal signals and no distal run off
* Infected Diabetic foot (DF) affecting heel and calf muscle with preserved knee joint
* Traumatic gangrene

Exclusion Criteria:

* Venous gangrene

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Wound healing rate | One year
  Rates of healing of different amputees
Incidence of infection | One year

SECONDARY OUTCOMES:
Function of the limb Rehabilitation Quality of life | Two years
  Incidence of recurrence
Mortality rate | Tow years

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mu Nagy, Study Director — Assiut University

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Kolossvary E, Farkas K, Karahan O, Golledge J, Schernthaner GH, Karplus T, Bernardo JJ, Marschang S, Abola MT, Heinzmann M, Edmonds M, Catalano M. The importance of socio-economic determinants of health in the care of patients with peripheral artery disease: A narrative review from VAS. Vasc Med. 2023 Jun;28(3):241-253. doi: 10.1177/1358863X231169316. Epub 2023 May 8. PMID 37154387
- [Background] Panhelleux B, Shalhoub J, Silverman AK, McGregor AH. A review of through-knee amputation. Vascular. 2022 Dec;30(6):1149-1159. doi: 10.1177/17085381211045183. Epub 2021 Nov 29. PMID 34844469
- [Background] Crane H, Boam G, Carradice D, Vanicek N, Twiddy M, Smith GE. Through-knee versus above-knee amputation for vascular and non-vascular major lower limb amputations. Cochrane Database Syst Rev. 2021 Dec 14;12(12):CD013839. doi: 10.1002/14651858.CD013839.pub2. PMID 34904714
- [Background] Howard RR, Chamberlain J, Macpherson AI. Through-knee amputation in peripheral vascular disease. Lancet. 1969 Aug 2;2(7614):240-2. doi: 10.1016/s0140-6736(69)90007-5. No abstract available. PMID 4184110
- [Background] Cull DL, Taylor SM, Hamontree SE, Langan EM, Snyder BA, Sullivan TM, Youkey JR. A reappraisal of a modified through-knee amputation in patients with peripheral vascular disease. Am J Surg. 2001 Jul;182(1):44-8. doi: 10.1016/s0002-9610(01)00663-8. PMID 11532414